CLINICAL TRIAL: NCT03643679
Title: Tobacco Cessation for Sexual Minorities
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 quarantines and closures prevented recruitment and assessment of participants.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kar-Hai Chu, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO18050656
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kwit smartphone app (Experimental): This arm will receive the Kwit smartphone app.
  Interventions: Other: Kwit smartphone app

INTERVENTIONS:
Other: Kwit smartphone app — The Kwit smartphone app combines several popular features of tobacco cessation apps, including game-like features (e.g., unlocking achievement milestones for completing cessation-related tasks), useful statistics (e.g., money saved), and an ability to share progress with friends. Users can actively engage with the app to track cravings or view progress, such as life expectancy gained. A passive component notifies users when milestones have been achieved, e.g., when blood no longer contains nicotine. Motivational messages can be actively requested at any time; they can also appear unsolicited, as when the user logs cravings.

SUMMARY:
There is a growing body of evidence revealing disproportionately higher rates of tobacco use among sexual and gender minority (SGM) individuals, compared to their heterosexual peers. These disparities have led organizations to support the inclusion of SGM in all local, state, and national tobacco prevention and control activities. In an attempt to leverage the online milieu for health-related interventions, mobile apps have been created to support tobacco cessation. However, evidence-based apps promoted by the National Cancer Institute are unpopular, remain poorly supported, and were not studied for use by SGM persons. Commercial apps, on the other hand, have been downloaded millions of times, contain many valuable features, and enjoy better infrastructure. Unfortunately, they are not evidence-based and have not been rigorously tested.

The University of Pittsburgh (Pitt) is currently conducting a randomized controlled trial to assess the feasibility and efficacy of using the Kwit tobacco cessation app with patients at UPMC Montefiore and Presbyterian hospitals (PI: Chu). It is a pragmatic clinical trial applying a patient-centered outcomes framework to ensure that-rather than focusing only on successful cessation-the study includes measurements for quality of life, mobility, and social interactions. We propose to extend the study to underrepresented SGM young adults.

Survey measures will be adapted as needed to address issues specific to the SGM population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Self-identified as a sexual minority (gay, lesbian, bisexual)
* Smokers interested in cessation (>1 cigarettes/day over the past 30 days)
* Must own an Apple or Android based smartphone.

Exclusion Criteria:

* Already receiving pharmacological and/or behavioral intervention or counseling for smoking cessation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Helpfulness, frequency of use, and ease of use of the intervention smartphone app | 1-month and 3-month
  Assessment of feasibility: Two follow-up surveys will be administered: the first, 1-month after recruitment,and the second, 3 months after recruitment. Surveys will be administered in-person. Specific questions will be asked to rate the Kwit smartphone application's feasibility, based on a combination of helpfulness, frequency of use, and ease of use. Frustrations and helpful aspects of the application will be assesses qualitatively.
  1. How helpful was the Kwit app?
  2. Was the app easy to use?
  3. Was it frustrating to use?
     Responses for 1-3 will be limited to Very helpful, Somewhat helpful, Neutral, Not very helpful, Not at all helpful
  4. What, if anything, was helpful about the app? What, if anything, was not helpful about the app?
  Each of these responses (Q1-3) will be combined to report a single overall feasibility value. Qualitative data (Q4) will be used to modify scores as needed.

SECONDARY OUTCOMES:
Cessation (self-report) | 1-month and 3-month
  Descriptive statistics will be used to assess cessation outcomes. The information will be obtained via two follow-up surveys (1 month and 3 months after recruitment), with specific questions pertaining to the level of participant smoking as well as their confidence levels on maintaining cessation.
  1. Since you joined the study, have you smoked a cigarette (even a puff)?
  2. How soon after you joined the study did you smoke your first cigarette, even a puff?
  3. In the past 30 days, on how many days did you smoke (even a puff)?
  4. (On the days you smoked) how many cigarettes on average did you smoke (even a puff)?
  5. In the past 7 days, have you smoked a cigarette, even a puff?
  6. How confident are you that you will be able to stay quit?
  The overall assessment of cessation will be primarily based on the 7-day item.
Cessation (bio-chemical) | 1-month and 3-month
  Cessation will also be verified by a breath analysis monitor. The information will be obtained during each follow-up. Biochemical verification will be based on a 10 COppm cutoff to determine whether or not the participant has successfully quit tobacco.

CONTACTS AND LOCATIONS:
Overall Officials: Kar-Hai Chu, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States